CLINICAL TRIAL: NCT07225192
Title: Therapy and Tech Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sean D Young, Professor of Emergency Medicine and Informatics, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00000488; 4R33AT010606 (NIH)
Record Dates: First submitted 2025-11-03; First posted 2025-11-06 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Generalized Anxiety Disorder (GAD); Major Depressive Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot Therapy Group (Experimental): Group 1 will be asked to use an AI chatbot like chatgpt as an adjunct to their regular therapy
  Interventions: Behavioral: Chatbot Therapy
- Control (No Intervention): Group 2 will be asked to continue their regular therapy as usual.

INTERVENTIONS:
Behavioral: Chatbot Therapy — This group will be asked to use an AI chatbot like chatgpt as an adjunct to their regular therapy
  Arms: Chatbot Therapy Group

SUMMARY:
The investigators want to test if gen AI can support therapy by recruiting patients already in therapy.

DETAILED DESCRIPTION:
Recent advancements in AI have led to chatbots, such as ChatGPT, capable of providing therapeutic responses. Early research evaluating chatbots' ability to provide relationship advice and single-session relationship interventions has showed that both laypeople and relationship therapists rate them high on attributes such as empathy and helpfulness. The investigators want to test if chatbots can be a good adjunct to traditional therapy. The investigators hypothesize that participants who regularly use a chatbot as an adjunct to traditional therapy will have better mental health outcomes. Participants will complete baseline, 4-week (post-intervention) and 4-week post-intervention measures and will be invited to gain their therapists ratings.

ELIGIBILITY:
Inclusion Criteria:

* 18+
* US Resident
* English-speaking
* Self-report having been treated for or diagnosed with generalized anxiety disorder or major depressive disorder by a licensed provider (e.g., MD, DO, LPCC, LCSW, LMFT) in the past 12 months
* Self-report currently being in individual therapy

Exclusion Criteria:

* Ever diagnosed with schizophrenia, schizoaffective disorder, bipolar disorder, or hospitalized for suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder (GAD-7) | Baseline, 4-week follow-up, 8-week follow-up
  Questions about symptoms of generalized anxiety disorder. Scale is 0-21. Higher scores is a worse outcome.
Patient Health Questionnaire (PHQ-9) | Baseline, 4-week follow-up, 8-week follow-up
  Questions about symptoms of depression. Scale is 0-27. Higher score is a worse outcome.

IPD SHARING:
Plan to Share IPD: No